CLINICAL TRIAL: NCT04212364
Title: An Evaluation of a Social Network Intervention for Primary and Secondary Prevention of Opioid Overdoses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 1R01CE003021 (NIH)
Record Dates: First submitted 2019-08-27; First posted 2019-12-27 (Actual); Last update posted 2024-01-24 (Actual); Status verified 2024-01

CONDITIONS: Overdose
Keywords: peer education; social networks
MeSH Terms: conditions — Drug Overdose

STUDY DESIGN:
Intervention Model Description: Index participants will be randomized into 1 of two study arms.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Peer Education (Experimental): * During Session 1, participants will be trained in Peer Education and how to use Nasal Narcan. They will be given two Nasal Narcan kit that includes 2 doses. One kit if for their use and one kit is to give someone in their social network after they have trained them in how to use it.
  * A week after Session 1, participants will be scheduled for Session 2.
  * During session 1 and 2 participants, Index participants will be taught information and skills pertaining to overdose prevention and response and how to train network members in overdose prevention and response.
  * At the 2nd session, index participants will be given 1 coupon to give to 1 member from their social network to attend Session 3.
  * Session 3 will be a dyad session where Index participants will use their peer mentors' skills to train their network member in overdose prevention and response.
  * Index participants will also be invited to up to 3 Booster Session (monthly) after they complete Sessions 1-3.
  Interventions: Behavioral: Peer Education; Drug: Narcan Nasal Product
- Standard of care (Active Comparator): * Participants randomized to this condition will participate in one 1-hour session. This session will be an individual session where the participant will meet with a trained staff member in a private room at the Lighthouse.
  * This session will be standard overdose prevention and response information. Participants will also be trained in Narcan administration. Participants will be given 1 nasal Narcan kit.
  * At the end of this session, participants will be asked to refer a network member to the study for survey visits
  Interventions: Drug: Narcan Nasal Product

INTERVENTIONS:
Behavioral: Peer Education — In this intervention, people who use opiates will be trained to be peer educators.
  Other Names: Experimental arm
  Arms: Peer Education
Drug: Narcan Nasal Product — All study participants will be trained in how to use nasal Narcan and they will receive a nasal Narcan kit.

SUMMARY:
The purpose of this study is to pilot and implement a peer mentor intervention focused on overdose prevention and care.

The intervention consists of 3 sessions. During the first and second session, each participant will meet individually with a trained staff member. In the 3rd session, the participant will invite a social network member to attend the session, and these 2 participants will meet with a trained staff member.

DETAILED DESCRIPTION:
The specific aims of the study are:

1. Conduct a pilot of an HIV/HCV/overdose prevention and care intervention for people who use opiates.
2. Evaluate the feasibility of collecting donated drug preparation containers (i.e., cookers) to assess the presence of fentanyl, HCV, and HIV.
3. Conduct a randomized controlled trial to assess efficacy of the experimental Peer Mentor condition on (a) overdose prevention and care education to drug network members, (b) naloxone availability, and (c) drug treatment readiness and entry.

There are two types of participants: Index participants and network participants. Both type of participant will currently used opiates. Participants will take part in a baseline visit and up to 3 follow-up visits. Index participants will be randomized into the intervention or control arm of the study.

ELIGIBILITY:
Inclusion Criteria for Index participants:

* self-reported use of opiates including heroin, fentanyl, or prescription opiates to get high at least 2 times in the last two weeks;
* willing to invite a network member who uses drugs to the study;
* ages 18-years or older;
* living in the Baltimore metropolitan region, and
* not previously enrolled in the study or currently enrolled in another Lighthouse study.

Inclusion Criteria for network participants:

* self-reported use of illicit injecting or non-injecting opiates at least 2 times in the last two weeks;
* sees the Index participant 2 or more times in the past week;
* ages 18 years or older; and
* living in the Baltimore metropolitan region.

Exclusion Criteria:

* Index participants may not take part in the study as a Network participant.
* Network participants may not take part in the study as an Index participant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 614 (Actual)
Dates: Start 2019-03-15 (Actual); Primary Completion 2023-12-29 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Network Enrollment | 6 months
  The question will be: How many people in their social network did Index participants recruit to the study? Participants provide a number of 0 or higher.

SECONDARY OUTCOMES:
Drug treatment entry | 12 months
  The question will be: In the past 12 months, did you enroll in a drug treatment program including a medically assisted treatment program? The response options are yes and no.
Overdose Risk | 12 months
  Change in risk will be measured by a score that includes frequency of naloxone availability when using opiates, testing drugs before injecting, and drug use alone. Higher scores will indicate increased overdose risk. Scores will be measured from 0-9

CONTACTS AND LOCATIONS:
Overall Officials: Carl A. Latkin, PhD, Principal Investigator — Johns Hopkins Bloomberg School of Public Health
Locations (1):
- Lighthouse Studies at Peer Point, Baltimore, Maryland, United States